CLINICAL TRIAL: NCT01772901
Title: A Randomized Controlled Trial of a Brief Educational Intervention to Increase Uptake of Influenza Vaccine Among Pregnant Women
Brief Title: Brief Influenza Vaccine Education to Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Marie Tarrant, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIV-INT-1
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Influenza; Infectious Disease; Pregnancy
Keywords: influenza; influenza vaccines; infectious disease; pregnancy
MeSH Terms: conditions — Influenza, Human; Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Usual outpatient antenatal care consists of routine checking of the maternal and foetal health by either clinic midwives or obstetricians along with health education to promote a healthy pregnancy.
- Influenza Vaccine Intervention (Experimental): The intervention group will receive a brief 5 to 10-minute educational talk by research nurse explaining the facts of influenza and influenza vaccine and answering participant questions.
  Interventions: Other: Influenza Vaccine Intervention

INTERVENTIONS:
Other: Influenza Vaccine Intervention — The intervention will include a brief 5 to 10-minute educational talk by research nurse explaining the facts of influenza and influenza vaccine and answering participant questions. The educational intervention will focus on: (1) Hong Kong government's recommendation regarding influenza vaccine during pregnancy, (2) potential complications associated with influenza during pregnancy and for young infants, (3) safety of influenza vaccine for mother and foetus, and (4) potential benefits of influenza vaccine for mother and infant, and (5) where and how to get the influenza vaccine in Hong Kong.
  Arms: Influenza Vaccine Intervention

SUMMARY:
The investigators will conduct a brief educational intervention to pregnant women who have not yet received the influenza vaccine in this pregnancy to improve the uptake of seasonal influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* 18 years of age or older
* in at least the second trimester of pregnancy
* Cantonese speaking
* Hong Kong resident
* no serious medical or obstetrical complications
* have not yet received the influenza vaccine in this pregnancy
* staying in Hong Kong for at least two weeks after delivery.

Exclusion Criteria:

* not entitled to health benefits in Hong Kong (NEP)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The proportion of influenza vaccination | 2 weeks postpartum
  The proportion of influenza vaccination in the control and intervention groups

SECONDARY OUTCOMES:
The influenza and influenza vaccine knowledge of participants | 2 weeks postpartum
  The influenza and influenza vaccine knowledge of participants in the control and intervention groups after receiving the intervention.
the proportion of participants initiating discussion about influenza vaccine with their health care provider | 2 weeks postpartum
the proportion of participants seeking out influenza vaccine | 2 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Marie TARRANT, PhD, MPH, RN, Principal Investigator — The University of Hong Kong
Locations (4):
- Hong Kong (4):
  - Kwong Wah Hospital, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tsan Yuk Hospital, Hong Kong

REFERENCES:
- [Derived] Wong VWY, Fong DYT, Lok KYW, Wong JYH, Sing C, Choi AY, Yuen CYS, Tarrant M. Brief education to promote maternal influenza vaccine uptake: A randomized controlled trial. Vaccine. 2016 Oct 17;34(44):5243-5250. doi: 10.1016/j.vaccine.2016.09.019. Epub 2016 Sep 22. PMID 27667330
- [Derived] Wong VW, Fong DY, Tarrant M. Brief education to increase uptake of influenza vaccine among pregnant women: a study protocol for a randomized controlled trial. BMC Pregnancy Childbirth. 2014 Jan 14;14:19. doi: 10.1186/1471-2393-14-19. PMID 24423245